CLINICAL TRIAL: NCT01290237
Title: The Use of a Loading Dose of Intravenous Vancomycin Will Achieve Therapeutic Concentration Earlier Than Conventional Pediatric Dosing: A Randomized Controlled Trial
Brief Title: Use of a Loading Dose of Vancomycin in Pediatric Dosing
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI leaving institution, slow enrollment
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Alicia Demirjian, Clinical Fellow, Pediatric Infectious Diseases, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10-11-0561
Record Dates: First submitted 2011-01-28; First posted 2011-02-04 (Estimated); Results first posted 2018-03-05 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-05

CONDITIONS: Infection
Keywords: vancomycin; loading dose; pharmacokinetic; pediatric; Methicillin-Resistant Staphylococcus aureus (MRSA); Serious infection with Gram positive bacteria
MeSH Terms: conditions — Infections | interventions — Vancomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vancomycin loading dose (Experimental): Intervention: administer intravenous vancomycin 30 mg/kg/dose once, followed 8 hours later by 20 mg/kg/dose every 8 hours
  Interventions: Drug: vancomycin hydrocloride
- Control (Active Comparator): No intervention. Administer intravenous vancomycin 20 mg/kg/dose every 8 hours as per hospital guideline.
  Interventions: Drug: vancomycin hydrocloride

INTERVENTIONS:
Drug: vancomycin hydrocloride — see description of study arms
  Other Names: Vancomycin

SUMMARY:
Vancomycin is an antibiotic administered to children or adults for many types of infections. While it has been used to treat infections of children for more than 50 years we are still not completely certain about the best dose to use when starting treatment with this medication.

This study is intended to evaluate whether giving a new higher dose of vancomycin for the first dose will help us get to the desired amount in the body more quickly then the usual first dose. Half of the patients would get the new higher dose and the other half of patients will get the typical first dose. Only the first dose is changed and all doses that follow are the same in both groups and are doses typically used for children.

DETAILED DESCRIPTION:
Setting and Patients We conducted a double-blind randomized controlled trial of children aged 2 to 18 years hospitalized at Boston Children's Hospital between February 1, 2011, and January 15, 2012, who required antimicrobial therapy with vancomycin (Hospira, Inc., Lake Forest, IL, lot #896188EO-4) for a suspected or documented infection. We excluded patients with a body weight above 67 kg (to limit the maximum loading dose to 2 g), preexisting severe renal dysfunction, defined as creatinine clearance <50 mL/min/1.73m2 using the original Schwartz equation,7 known hearing impairment, intravenous vancomycin treatment in the prior 7 days or undergoing a procedure with anticipated moderate to severe blood loss (eg, cardiac surgery or extensive orthopedic procedure).

For all participants enrolled in the study, relevant baseline demographic, medical history and safety data were recorded. Medical history data included primary and secondary diagnoses; other comorbidities such as obesity or cystic fibrosis; and presence of systemic inflammatory response syndrome, defined as 2 or more of the following: temperature >38.5°C or <36°C; mean heart rate >2 standard deviations above normal for age; mean respiratory rate >2 standard deviations above normal for age; or high or low white blood cell count for age.

Randomization and Concealment Participants were randomized in blocks of 2 and 4 to receive either a loading dose of 30 mg/kg of vancomycin as a single intravenous infusion over 2 hours (intervention group) or an initial vancomycin dose of 20 mg/kg intravenously over 2 hours (comparison group). The initial dose was administered over 2 hours in both groups to preserve allocation concealment. All patients subsequently received a 20 mg/kg dose every 8 hours as was the standard of care in our hospital for treatment of severe infections at the time of the study. Subsequent doses were administered over 1 hour, unless the patient developed red man syndrome (as identified by the clinical team), in which case the infusion time was increased to 2 hours. The investigators, family and primary care teams were blinded to group assignment, and the first dose of vancomycin for all participants was prepared so that the solution volumes were identical. The computer-generated randomization was concealed in a locked binder until the intervention was assigned.

Vancomycin Concentration Sampling and Analysis Trough serum vancomycin concentrations were obtained within 60 minutes before the second (8-hour) and third (16-hour) vancomycin doses. In order to increase the likelihood of having a cloud of sparse data for population pharmacokinetic analysis, 1 or 2 additional serum vancomycin samples were obtained from each participant within the first 32 hours of therapy at a time coinciding with blood collection for clinical care. These samples were obtained only from participants with an indwelling catheter whose family provided written consent for additional sampling.

Vancomycin concentrations were measured using a fluorescence polarization immunoassay (Roche Diagnostics, Indianapolis, IN) on the Roche Integra 800 instrument. The assay had a limit of quantitation of 0.74 mg/L and an interassay coefficient of variability of <3%.

ELIGIBILITY:
Inclusion Criteria:

* Receiving care at Children's Hospital Boston
* Prescribed intravenous vancomycin by their physician

Exclusion Criteria:

* Weight above 67 kg
* Pre-existing renal dysfunction (creatinine clearance < 50 ml/min/1.73m2)
* Known hearing impairment
* Recent intravenous vancomycin treatment (within 7 days)
* Undergoing procedure with anticipated moderate-severe blood loss

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 59 (Actual)
Dates: Start 2011-02; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alicia A Demirjian, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

REFERENCES:
- [Background] Rybak M, Lomaestro B, Rotschafer JC, Moellering R Jr, Craig W, Billeter M, Dalovisio JR, Levine DP. Therapeutic monitoring of vancomycin in adult patients: a consensus review of the American Society of Health-System Pharmacists, the Infectious Diseases Society of America, and the Society of Infectious Diseases Pharmacists. Am J Health Syst Pharm. 2009 Jan 1;66(1):82-98. doi: 10.2146/ajhp080434. No abstract available. PMID 19106348
- [Background] Frymoyer A, Hersh AL, Benet LZ, Guglielmo BJ. Current recommended dosing of vancomycin for children with invasive methicillin-resistant Staphylococcus aureus infections is inadequate. Pediatr Infect Dis J. 2009 May;28(5):398-402. doi: 10.1097/INF.0b013e3181906e40. PMID 19295465
- [Background] Liu C, Bayer A, Cosgrove SE, Daum RS, Fridkin SK, Gorwitz RJ, Kaplan SL, Karchmer AW, Levine DP, Murray BE, J Rybak M, Talan DA, Chambers HF; Infectious Diseases Society of America. Clinical practice guidelines by the infectious diseases society of america for the treatment of methicillin-resistant Staphylococcus aureus infections in adults and children. Clin Infect Dis. 2011 Feb 1;52(3):e18-55. doi: 10.1093/cid/ciq146. Epub 2011 Jan 4. PMID 21208910
- [Derived] Demirjian A, Finkelstein Y, Nava-Ocampo A, Arnold A, Jones S, Monuteaux M, Sandora TJ, Patterson A, Harper MB. A randomized controlled trial of a vancomycin loading dose in children. Pediatr Infect Dis J. 2013 Nov;32(11):1217-23. doi: 10.1097/INF.0b013e3182a26774. PMID 23817340

RESULTS

PARTICIPANT FLOW:
Groups:
- Vancomycin Loading Dose: Intravenous vancomycin 30 mg/kg/dose once, followed 8 hours later by 20 mg/kg/dose every 8 hours
  intravenous vancomycin hydrochloride: see description of study arms
- Control: Intravenous vancomycin 20 mg/kg/dose every 8 hours
  intravenous vancomycin hydrochloride: see description of study arms
Period: Overall Study
Arm/Group | Vancomycin Loading Dose | Control
Started | 30 | 29
Completed | 19 | 27
Not Completed | 11 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vancomycin Loading Dose | Control | Total
Number analyzed (Participants) | 30 | 29 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.63 (4.4) | 8.76 (4.04) | 8.70 (4.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 15 | 27
  Male | 18 | 14 | 32
Region of Enrollment [Number; unit: participants]
  United States | 30 | 29 | 59

OUTCOME MEASURES:

1. Primary Outcome: Count of Participants With Vancomycin Trough Between 15 and 20
Description: proportion of participants whose vancomycin trough was between 15 and 20 mcg/mL, 8 hours after the first vancomycin dose, in loading dose group as compared to control group
Time Frame: 8 hours after the first dose of vancomycin
Population: Loading dose - trough at 8 hours was not collected for 11 participants: vancomycin was discontinued prior to second dose (7), participant changed their mind (1), other reason (3) Among participants allocated to conventional treatment, trough at 8 hours was not collected for 2: vancomycin discontinued prior to second dose (1), changed mind (1)
Measure: Count of Participants; unit: Participants
Arm/Group | Vancomycin Loading Dose | Control
Number analyzed (Participants) | 19 | 27
Participants | 2 | 0

2. Secondary Outcome: AUC/MIC for Vancomycin in the Study Population
Description: AUC/MIC using hypothetical MIC = 1 mg/L
Time Frame: within 48 hours after receiving the first dose of vancomycin
Population: Number of measurements reflects the number of participants with blood samples available for testing
Measure: Mean (Standard Deviation); unit: AUC/MIC ratio
Groups:
- Loading Dose; Conventional Dose: As above
Arm/Group | Loading Dose | Conventional Dose
Number analyzed (Participants) | 25 | 26
AUC/MIC ratio | 446.5 (195.5) | 434.0 (153.2)

ADVERSE EVENTS:
Arm/Group | Vancomycin Loading Dose | Control
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/29
Serious Adverse Events (participants affected / at risk) | 1/30 | 0/29
Other Adverse Events (participants affected / at risk) | 20/30 | 11/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vancomycin Loading Dose (N=30) | Control (N=29)
acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) — One patient with cystic fibrosis developed acute kidney injury 7 days after administration of a conventional dose while receiving concomitant nephrotoxic medications; renal function recovered when these medications and vancomycin were discontinued.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vancomycin Loading Dose (N=30) | Control (N=29)
Red man syndrome (Skin and subcutaneous tissue disorders) | 14 (14) | 7 (7)
Escalation of care within 7 days (General disorders) | 2 (2) | 3 (3)
Doubling of baseline creatinine (Renal and urinary disorders) | 4 (4) | 1 (1)

LIMITATIONS AND CAVEATS:
* trial underpowered to detect an increase of ≥40% in concentrations (small sample size)
* more cases excluded in the high-dose group than in reference group (possible analysis bias)
* increase in red man syndrome in the high-dose group

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No